CLINICAL TRIAL: NCT02034487
Title: Delayed Puberty in Boys; Clinical and Biochemical Characteristics and Effect of Testosterone Treatment - Retrospective Experience From a Single Tertiary Referral Centre 1990-2013
Brief Title: Delayed Puberty in Boys; Clinical and Biochemical Characteristics and Effect of Testosterone Treatment
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, PhD, DMSc, Rigshospitalet, Denmark
Other Study IDs: KF01328087
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Delayed Puberty
Keywords: Delayed Puberty; Boys; Hormones; Polymorphism, Genetic
MeSH Terms: conditions — Puberty, Delayed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum and white cells

GROUPS / COHORTS (1):
- Boys with delayed puberty: Boys with no signs of puberty by an age that is -2 standard deviation below the population mean.
  Interventions: Other: retrospective data collection

INTERVENTIONS:
Other: retrospective data collection

SUMMARY:
To evaluate the phenotype and biochemical characteristics of boys referred for delayed puberty, to describe the frequency of associated co-morbidities and diseases, to evaluate the diagnostic criteria and the effect of testosterone treatment.

DETAILED DESCRIPTION:
Delayed Puberty in Boys; Clinical and biochemical characteristics and effect of testosterone treatment, is a retrospective study in a large case series of Danish boys with delayed puberty.

All boys were referred to the Department of Growth and Reproduction to be evaluated for delayed puberty.

Medical history: Birth length, birth weight, gestational age at birth, medical history (including cryptorchidism and hypospadias), family history of delayed puberty in mother, father and possible siblings.

Physical examination: Pubertal staging according to Tanners classification of boys, genitalia development (G1-G5), pubic hair development (PH1-PH6), axillary hair (yes/no), axillary sweat (yes/no), gynecomastia (yes/no), micropenis (yes/no), height, mother height, father height, target height, weight, BMI, bone age and predicted adult height.

Blood sampling for measurement of hormone levels: Follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol, anti-mullerian hormone, sex hormone-binding globulin, testosterone, dehydroepiandrosterone-sulfate, androstenedione, inhibin A, inhibin B, growth hormone, insulin like growth factor-1 and insulin like growth factor binding protein-3.

Gonadotropin-releasing hormone stimulation test for measurement of peak FSH and peak LH.

Retrospective DNA analysis looking for common polymorphisms.

If testosterone treatment were initiated, route of administration, dose and duration of treatment were registered.

ELIGIBILITY:
Inclusion Criteria:

* All boys identified in the period from January 1990 to February 2013

Exclusion Criteria:

* Misclassified (other diagnoses)
* Insufficient data
* Lost to follow up

Ages: 13 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of boys who were referred to be evaluated for delayed puberty at the Department of Growth and Reproduction between January 1990 and February 2013.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 1990-01; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Age at diagnosis in boys with delayed puberty. | At first evaluation
  We will evaluate the mean age at diagnosis as well as the age distribution of newly diagnosed boys. These data are compared to age at onset and progression of normal puberty in contemporary healthy Danish boys.

SECONDARY OUTCOMES:
Selected secondary outcomes include clinical, auxological and biochemical parameters and association to specific genetic polymorphisms | At first evaluation and during first 12 months of observation / treatment
  Specifically, genital stage, pubic hair stage, axillary hair, axillary sweat, gynecomastia, micropenis, height, mother height, father height, target height, weight, BMI, bone age and predicted adult height. We will evaluate serum levels of follicle stimulating hormone, luteinizing hormone, estradiol, anti-mullerian hormone, sex hormone-binding globulin, testosterone, dehydroepiandrosterone-sulfate, androstenedione, inhibin A, inhibin B, growth hormone, insulin like growth factor-1 and insulin like growth factor binding protein-3. We will evaluate the effect of candidate polymorphisms suspected to affect pubertal timing, e.g. FSHR, FSHB, FGF23, KISS1, NeurokininB, GnRH, GnRH-R, LH, LH-R, GHRd3.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, PhD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Lawaetz JG, Hagen CP, Mieritz MG, Blomberg Jensen M, Petersen JH, Juul A. Evaluation of 451 Danish boys with delayed puberty: diagnostic use of a new puberty nomogram and effects of oral testosterone therapy. J Clin Endocrinol Metab. 2015 Apr;100(4):1376-85. doi: 10.1210/jc.2014-3631. Epub 2015 Jan 16. PMID 25594861